CLINICAL TRIAL: NCT02799355
Title: Treatment of Chronic Hepatitis With Sofosbuvir in Combination With Ribavirin With or Without Pegylated Interferon: North India Gastroenterology Consortium
Acronym: GCNI-CHC
Status: Completed | Type: Observational
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Professor, Dayanand Medical College and Hospital
Other Study IDs: GCNI-CHC
Record Dates: First submitted 2016-05-18; First posted 2016-06-14 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis, Chronic
MeSH Terms: conditions — Hepatitis, Chronic | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sofosbuvir, Ribavirin, With or Without Pegylated Interferon — Retrospective will carried out to find percentage of patients with sustained virologic response at 12 weeks after the end of treatment
  Other Names: Sofosbuvir in Combination With Ribavirin With or Without Pegylated Interferon

SUMMARY:
Of the six main genotypes of the hepatitis C virus (HCV), genotypes 2 and 3 account for approximately 30% of chronic infections worldwide. In North India, Genotypes 3 and 1 account for 95% of chronic hepatitis C patients The first three direct-acting antiviral agents to receive FDA approval-boceprevir, telaprevir, and simeprevir-do not currently have a role in the treatment of genotype 3 infection. In contrast, the direct-acting antiviral agents, daclatasvir and sofosbuvir, have good activity against all genotypes. The SVR rates of 90 - 100% in genotype 3 were achieved with oral sofosbuvir plus ribavirin regimen to 24 weeks. Similar SVR rates were achieved in Genotype 1 with oral sofosbuvir plus weight based ribavirin and Pegylated Interferon alpha 2 a. However, the ongoing discovery and development of agents that directly target various stages of HCV replication are likely to provide HCV-infected patients with effective interferon-free therapy. HCV genotype 3 infection is associated with a higher incidence of hepatic steatosis, more rapid progression of fibrosis, and possibly a greater risk of hepatocellular carcinoma than is HCV genotype 2 infection.Moreover, patients with HCV genotype 3 infection are less responsive to peginterferon based treatment than are patients with HCV genotype 2 infection.

DETAILED DESCRIPTION:
Sofosbuvir is an oral nucleotide analogue inhibitor of the HCV NS5B polymerase that is effective against HCV genotypes 2 and 3 when it is administered in combination with weight based ribavirin for 24 weeks. In Genotype 1, a combination of Pegylated Interferon alpha 2 a with oral Sofosbuvir and weight based Ribavirin for 12 weeks resulted in 90 -100 % sustained virological response rates (SVR). These SVR rates for chronic hepatitis C genotypes 1,2 and 3 are all based on Western studies. The investigators plan to conduct a retrospective study in Northern India region on patients treated with Sofosbuvir and Ribavirin or Sofosbuvir, Ribavirin and Peginterferon alpha 2a. The purpose of the investigators study is to assess the percentage of patients with sustained virologic response.

ELIGIBILITY:
Inclusion Criteria:

* Age more then 18 years.
* Patient who on treatment of either Sofosbuvir and Ribavirin (24 weeks) or Sofosbuvir, Ribavirin and peginterferon (12 weeks).

Exclusion Criteria:

* Patient who are lost to follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a retrospective study conducted on 1500 to 2000 patients who have recieved treatment of Sofosbuvir and Ribavirin or Sofosbuvir, Ribavirin and peg interferon alpha 2a
Sampling Method: Probability Sample
Enrollment: 1203 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sustained virologic response at 12 weeks after the end of treatment. | 3 month
  Sustained virologic response was defined as a level of HCV RNA below the lower limit of quantification (25 IU per milliliter)

SECONDARY OUTCOMES:
Side effect | 3 month
  Assess the treatment side effect

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, D.M.C. and Hospital, Ludhiana, Punjab, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tapper EB, Afdhal NH. Is 3 the new 1: perspectives on virology, natural history and treatment for hepatitis C genotype 3. J Viral Hepat. 2013 Oct;20(10):669-77. doi: 10.1111/jvh.12168. PMID 24010641
- [Result] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2011 Aug;55(2):245-64. doi: 10.1016/j.jhep.2011.02.023. Epub 2011 Mar 1. No abstract available. PMID 21371579
- [Result] Goossens N, Negro F. Is genotype 3 of the hepatitis C virus the new villain? Hepatology. 2014 Jun;59(6):2403-12. doi: 10.1002/hep.26905. Epub 2014 Apr 14. PMID 24155107
- [Result] Wartelle-Bladou C, Le Folgoc G, Bourliere M, Lecomte L. Hepatitis C therapy in non-genotype 1 patients: the near future. J Viral Hepat. 2012 Aug;19(8):525-36. doi: 10.1111/j.1365-2893.2012.01634.x. PMID 22762136
- [Result] Marcellin P, Cheinquer H, Curescu M, Dusheiko GM, Ferenci P, Horban A, Jensen D, Lengyel G, Mangia A, Ouzan D, Puoti M, Rodriguez-Torres M, Shiffman ML, Schmitz M, Tatsch F, Rizzetto M. High sustained virologic response rates in rapid virologic response patients in the large real-world PROPHESYS cohort confirm results from randomized clinical trials. Hepatology. 2012 Dec;56(6):2039-50. doi: 10.1002/hep.25892. Epub 2012 Aug 8. PMID 22706730
- [Result] Alberti A. Optimizing PEG-interferon and ribavirin combination therapy for patients infected with HCV-2 or HCV-3: is the puzzle completed? J Hepatol. 2004 Jun;40(6):1032-5. doi: 10.1016/j.jhep.2004.04.008. No abstract available. PMID 15158348
- [Result] Manns MP, von Hahn T. Novel therapies for hepatitis C - one pill fits all? Nat Rev Drug Discov. 2013 Aug;12(8):595-610. doi: 10.1038/nrd4050. Epub 2013 Jun 28. PMID 23807378
- [Result] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594
- [Result] Zeuzem S, Dusheiko GM, Salupere R, Mangia A, Flisiak R, Hyland RH, Illeperuma A, Svarovskaia E, Brainard DM, Symonds WT, Subramanian GM, McHutchison JG, Weiland O, Reesink HW, Ferenci P, Hezode C, Esteban R; VALENCE Investigators. Sofosbuvir and ribavirin in HCV genotypes 2 and 3. N Engl J Med. 2014 May 22;370(21):1993-2001. doi: 10.1056/NEJMoa1316145. Epub 2014 May 4. PMID 24795201
- [Result] Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Symonds WT, Hindes RG, Berrey MM. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med. 2013 Jan 3;368(1):34-44. doi: 10.1056/NEJMoa1208953. PMID 23281974
- [Result] Chakravarti A, Dogra G, Verma V, Srivastava AP. Distribution pattern of HCV genotypes & its association with viral load. Indian J Med Res. 2011 Mar;133(3):326-31. PMID 21441689
- [Result] Singh S, Malhotra V, Sarin SK. Distribution of hepatitis C virus genotypes in patients with chronic hepatitis C infection in India. Indian J Med Res. 2004 Apr;119(4):145-8. PMID 15147119